CLINICAL TRIAL: NCT04851418
Title: Pre-hOspital Evaluation of Chest Pain Patients With sUspected Non ST-segment eLevation myocARdial Infarction Using the HEART-score With a Troponin Point-of-care Test
Acronym: POPular HEART
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: St. Antonius Hospital (Other)
Collaborators: Diakonessenhuis, Utrecht (Other); Abbott (Industry)
Responsible Party: Principal Investigator, J.M. ten Berg, Prof. Dr. J.M. ten Berg, St. Antonius Hospital
Other Study IDs: NL71897.100.19
Record Dates: First submitted 2021-04-12; First posted 2021-04-20 (Actual); Last update posted 2021-04-20 (Actual); Status verified 2021-04

CONDITIONS: Coronary Artery Disease
Keywords: acute coronary syndrome; point of care troponin; HEART score; NSTE-ACS
MeSH Terms: conditions — Coronary Artery Disease; Acute Coronary Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — two venous blood samples will be drawn in the pre-hospital phase. One will be used for high-sensitive troponin measure in the pre-hospital phase (at the resident of the patient).
  The second one will be used to validate the point-of-care measurement with the troponin value in the laboratory.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- Possible NSTE-ACS: All patients with a suspicion of non-ST-elevation acute coronary syndrome (NSTE-ACS) in the pre-hospital phase are eligible for inclusion. In all included patients, the POC cTn will be performed and the HEART-score will be calculated in the pre-hospital phase. Simultaneously, a venous blood sample will be drawn from the venous access site for later hs-cTn testing. Outcomes of both the POC cTn or the pre-hospital HEART-score will be blinded for the physicians at the emergency department (ED) and will not affect current treatment strategy. All patients with suspected NSTE-ACS will undergo hs-cTn testing and the HEART-score will also be calculated at the ED (T1, standard of care). Here, an additional venous blood sample will be drawn next to routine blood testing testing (T1).
  Interventions: Device: Possible NSTE-ACS

INTERVENTIONS:
Device: Possible NSTE-ACS — As mentioned in the group description
  Other Names: Point of Care troponin I iSTAT Abbot

SUMMARY:
Overcrowding in the emergency department is an increasing problem in hospitals worldwide. Point-of-care Troponin (POC cTn) testing combined with a well investigated risk stratification tool (HEART-score) used in the ambulance may contribute to more rapidly diagnostics of ruling in or ruling out myocardial infarctions (MI) and subsequently reduce unnecessary hospital admissions, total admission time and costs. However, the applicability of the POC cTn and the HEART-score in the pre-hospital setting remains unclear. This study will evaluate this applicability.

DETAILED DESCRIPTION:
Co-primary Objectives:

1. To evaluate the interobserver agreement of the HEART-score performed by ambulance personnel compared to the HEART-score performed by emergency physicians.
2. To evaluate the diagnostic performance of a strategy based on a pre-hospital HEART-score (with POC cTn testing) or combined with an adjuvant single hs-cTn test at the emergency department to rule-in or rule-out acute coronary syndrome (ACS).
3. To evaluate the diagnostic performance of (serial) POC cTn testing or combined with hs-cTn testing compared to (serial) hs-cTn testing to rule-in or rule-out MI.
4. To investigate the feasibility of using the pre-hospital HEART-score and POC cTn in the 0/1 hour algorithm to rule-out ACS.

   Secondary Objectives:
5. To evaluate the occurrence of major adverse cardiac events (MACE) in all included patients with a follow up time of 30 days from first medical contact.
6. To evaluate the patient reported outcome measures (PROMs) in all chest pain patients transported to the hospital at baseline and at 30 days
7. To perform a cost-analysis of an early diagnostic strategy using the pre-hospital HEART-score

Study design: A prospective, observational, single multicentre study Study population: Total number of patients needed for analysis: n=650 Inclusion criteria: - All out-of-hospital chest pain patients visited by an ambulance

* Transportation to a hospital with working diagnosis NSTE-ACS
* Age ≥ 18 years Exclusion criteria: - Comatose state, hemodynamic instability or shock
* Electrocardiographic ST-segment elevation in the pre-hospital setting treated as STEMI
* No pre-hospital 12-lead electrocardiogram performed or available
* An obvious non-cardiac cause for the chest pain (trauma, etc.)
* Suspicion of aortic dissection or pulmonary embolism
* Cognitive impairment
* Pregnancy
* Suspicion of COVID-19 by ambulance

Study procedures: The HEART-score and the POC cTn will be calculated in all included patients in the pre-hospital phase. Simultaneously, a venous blood sample will be drawn from the venous access site for later hs-cTn testing. Outcomes of any pre-hospital study measurements (i.e. pre-hospital POC cTn results or calculated pre-hospital HEART-scores) are blinded to the physicians at the ED and will not affect usual care. According to current practice, all patients will be transported to the hospital for further evaluation. At the emergency department (ED) all included patients will undergo regular hs-cTn testing and HEART-score assessment performed by emergency physicians (standard care), and an extra venous blood sample will be drawn for this study. Additional cTn tests (POC and hs-cTn) will be performed in the laboratory.

Main study parameters/endpoints:

1. HEART-score agreement (interobserver variability between pre-hospital and in-hospital HEART-score assessment)
2. Final diagnosis of NSTE-ACS at discharge
3. Myocardial infarction at discharge

   Secondary study parameters/endpoints:
4. Composite endpoint (cardiovascular mortality, myocardial infarction, urgent revascularisation) at 30 days
5. Angina frequency and stability, physical limitations, treatment satisfaction, quality-of-life, cardiac anxiety and depression (SAQ, PHQ-4)

Follow-up: Total follow-up duration is 30 days after initial presentation. Other demographic and clinical parameters at baseline will be taken into account.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: All patients will undergo a POC cTn test performed by ambulance personnel. In all patients, two venous blood samples will be drawn in the pre-hospital phase (1x) and at the emergency department (1x). Besides the minimal risks of performing a POC finger prick test, no other risks are involved with study participation. All patients will be asked to fill in questionnaires (i.e. SAQ, PHQ-4) at baseline and at follow-up.

ELIGIBILITY:
Inclusion Criteria:

* All out-of-hospital chest pain patients visited by an ambulance
* Transportation to a hospital with working diagnosis NSTE-ACS
* Age ≥ 18 years

Exclusion Criteria:

* Comatose state, hemodynamic instability or shock
* Electrocardiographic ST-segment elevation in the pre-hospital setting
* No pre-hospital 12-lead electrocardiogram performed or available
* An obvious non-cardiac cause for the chest pain (trauma, etc.)
* Suspicion of aortic dissection or pulmonary embolism
* Cognitive impairment
* Pregnancy

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with suspected acute coronary syndrome. Total number of patients needed for analysis: n=650
Sampling Method: Probability Sample
Enrollment: 650 (Estimated)
Dates: Start 2020-09-01 (Actual); Primary Completion 2022-01 (Estimated); Study Completion 2022-02 (Estimated)

PRIMARY OUTCOMES:
Heart score agreement | 1 year
  HEART-score agreement (interobserver variability between pre-hospital and in-hospital HEART-score assessment): the calculated heart score by the ambulance will be subtracted from the calculated score of the emergency department. The minimum value could be -10 and the maximum value could be +10. A positive score means that the ambulance estimates the patient to be sicker or at higher risk. A negative value means that the ED estimates the patient to be sicker/at higher risk for developing major adverse cardiac events.
Number of participants with final diagnosis of NSTE-ACS | 1 year
  final diagnosis of NSTE-ACS (non-ST elevation myocardial infarction and unstable angina pectoris) at discharge
Number of participants with final diagnosis of myocardial infarction at discharge | 1 year
  Myocardial infarction at discharge

SECONDARY OUTCOMES:
Number of participants with a composite endpoint | 30 days
  4. The composite endpoint exists out of cardiovascular mortality, myocardial infarction, urgent revascularisation at 30 days
Patient reported outcome measure: Seattle Angina questionnaire (SAQ) | 30 days
  In order to gain information regarding how patients experience their disease, 2 questionnaires will be sent. The first questionnaire; Seattle Angina questionnaire will assess: angina frequency and stability, physical limitations, treatment satisfaction, and quality-of-life.
Patient reported outcome measure: Patient Health Questionnaire 4 | 30 days
  In order to gain information regarding how patients experience their disease, 2 questionnaires will be sent. The second questionnaire will be the Patient Health Questionnaire 4, will discuss topics such as anxiety, depression and general psychological distress.

CONTACTS AND LOCATIONS:
Overall Officials: HJ Houtgraaf, Dr., Principal Investigator — Diakonessenhuis, Utrecht
Locations (2):
- Netherlands (2):
  - St Antonius Hospital, Nieuwegein
  - Diakonessenhuis Utrecht, Utrecht

IPD SHARING:
Plan to Share IPD: No
nine

REFERENCES:
- [Derived] Azzahhafi J, Chan Pin Yin DR, Epping M, Bofarid H, Rikken SA, Verhagen T, Boomars R, Radstok A, Houtgraaf J, Bikker A, Ten Berg JM. Pre-hospital evaluation of chest pain patients using the modified HEART-score: rationale and design. Future Cardiol. 2024 Apr 25;20(5-6):241-250. doi: 10.1080/14796678.2024.2356995. Epub 2024 Jun 28. PMID 38940186